CLINICAL TRIAL: NCT02324062
Title: University of Southern California (USC) Norris Comprehensive Cancer Center and Stanford Cancer Institute Cancer Genetics Hereditary Cancer Panel Testing
Brief Title: Cancer Genetics Hereditary Cancer Panel Testing
Acronym: HCP
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 0S-13-1
Record Dates: First submitted 2014-12-14; First posted 2014-12-24 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Hereditary Breast and Ovarian Cancer
Keywords: Cancer Genetics; Multi-gene cancer panel testing
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Pathogenic group: Blood Draw and Baseline Questionnaire: Participants will have their blood drawn for the study and complete a baseline questionnaire about their current cancer screening practices and concern regarding cancer.
  Patients identified with a mutation in a gene not commonly tested for prior to the advent of multiplex panel testing. This excludes BRCA1, BRCA2, MLH1, MSH2, MSH6, PMS2, EPCAM, APC, MYH unless a patient tested positive for one of these 9 genes but did not meet clinical criteria for the underlying syndrome (n = 124). These participants will be asked to complete questionnaires for the duration of the study (up to 60 months after enrollment) at 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months.
  Interventions: Other: Questionnaires; Other: Blood Draw and Baseline Questionnaire
- VUS group: Blood Draw and Baseline Questionnaire: Participants will have their blood drawn for the study and complete a baseline questionnaire about their current cancer screening practices and concern regarding cancer.
  Patients identified with a variant of unknown significance of any gene of any nonBRCA (BRCA1 and BRCA2) or non-Lynch syndrome gene (MLH1, MSH2, MSH6, PMS2 and EPCAM).
  Target accrual is 100. These participants will be asked to complete questionnaires for the duration of the study (up to 60 months after enrollment) at 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months.
  Interventions: Other: Questionnaires; Other: Blood Draw and Baseline Questionnaire
- Negative Group: Blood Draw and Baseline Questionnaire: Participants will have their blood drawn for the study and complete a baseline questionnaire about their current cancer screening practices and concern regarding cancer.
  Patients who test negative for all the genes tested. Target goal is 50 for Stanford (100 for the study). These participants will be asked to complete questionnaires for the duration of the study (up to 60 months after enrollment) at 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months.
  Interventions: Other: Questionnaires; Other: Blood Draw and Baseline Questionnaire
- No follow-up intervention group: Blood Draw and Baseline Questionnaire: Participants will have their blood drawn for the study and complete a baseline questionnaire about their current cancer screening practices and concern regarding cancer.
  All other participants who do not meet any of the above criteria or fall into one of these groups after the target goal is met for that group.
  Interventions: Other: Blood Draw and Baseline Questionnaire

INTERVENTIONS:
Other: Questionnaires — These participants will be asked to complete questionnaires for the duration of the study (up to 60 months after enrollment) at 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months.
  Groups: Negative Group; Pathogenic group; VUS group
Other: Blood Draw and Baseline Questionnaire — Participants will have their blood drawn for the study and complete a baseline questionnaire about their current cancer screening practices and concern regarding cancer.

SUMMARY:
This study is about understanding the use of a genetic test (Myriad Genetics myRisk panel) that analyzes 25 genes related to different hereditary cancer conditions. The investigators hope to learn more about how this type of genetic test is used clinically. The investigators also hope to understand more about the experience of individuals and families who undergoing this test of genetic testing.

DETAILED DESCRIPTION:
If a patient is identified as fulfilling one of the screening criteria, possible participants should be referred to the Cancer Genetics Clinic for further evaluation for possible enrollment into the study. A pre-clinic questionnaire will be sent to the patients prior to their assessment in cancer genetics clinic in order to obtain baseline information that will be used to inform changes during follow-up. Assessments performed exclusively to determine eligibility for this study will be done only after obtaining informed consent. Assessments performed for clinical indications (not exclusively to determine study eligibility) may be used for baseline values even if the studies were done before informed consent was obtained.

All screening procedures must be performed on the day of registration unless otherwise stated. The screening procedures include:

1. Medical history -Complete medical and surgical history, family history including a multi-generation family pedigree, and social history
2. Demographics - Age, gender, race, ethnicity
3. Review subject eligibility criteria
4. Physical exam including vital signs, height and weight
5. Blood draw for correlative studies
6. DNA from whole blood will be isolated

Intervention Procedure:

Approximately 15 ml of blood will be drawn at the time of enrollment (one time blood draw) and sent to Myriad Genetics and Laboratories for analysis of 25 genes using next generation sequencing. This platform will sequence 25 genes in one experimental run and the results will be sent back to the cancer genetics clinic for interpretation and disclosure.

Randomization of the patient Population:

After results are given to the patient they will be randomized into 4 groups:

* Patients identified with a mutation in a gene not commonly tested for prior to the advent of multiplex panel testing. This excludes BRCA1, BRCA2, MLH1, MSH2, MSH6, PMS2, EPCAM, APC, MYH unless a patient tested positive for one of these 9 genes but did not meet clinical criteria for the underlying syndrome (Stanford accrual goal is 62/USC 62)
* Patients identified with a variant of unknown significance (VUS) of any gene of any nonBRCA (BRCA1 and BRCA2) or non-Lynch syndrome gene (MLH1, MSH2, MSH6, PMS2 and EPCAM).

Stanford target accrual is 50 and 50 for USC.

* Patients who test negative for all the genes tested. Target goal is 50 for Stanford/50 for USC for the study.
* All other participants who do not meet any of the above criteria or fall into one of these groups after the target goal is met for that group. Only participants who are in the 1st three groups will be asked to complete questionnaires for the duration of the study (up to 60 months after enrollment)

Follow-up Procedures:

Patients (as noted above) will be followed at 3 months, 6 months, 12 months, 24 months, 36 months, 48 months, and 60 months

• At 3 months and 6 months after disclosure of genetic testing results, follow up questionnaires will ask if participants had initiated or intend to undergo any of the following risk reducing interventions and/or treatment: (i) Cancer surveillance/screening: breast MRI, mammograms, self-breast examinations, thyroid ultrasound, dermatology exams, urinalysis, upper endoscopy, colonoscopy, endometrial biopsy, transvaginal ultrasound, or other imaging (i.e. whole body rapid MRI) (ii) Chemoprevention/Behavior Modification: Tamoxifen, Oral Contraceptives (OCP), Raloxifene, Sulindac, Abstinence from Smoking (iii) Prophylactic procedures: Mastectomy, TAHBSO, polypectomy, total and segmental colectomy (iv) Cancer Treatment: aggregated pharmacologic and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:Screening Criteria Patients meeting one of the following criteria will be eligible for screening the study.

* Any individual with multiple primary cancers
* Any individual diagnosed with cancer under age 50
* Individuals with two or more first or second-degree relatives with cancer.
* Individuals from families where at least one family member was diagnosed with cancer under age 50
* Individuals meeting a phenotypic diagnosis of specific hereditary cancer syndromes including, but not limited to:

  * Hereditary Breast and Ovarian Cancer
  * Lynch Syndrome
  * Familial or Attenuated Adenomatous Polyposis Syndrome
  * Hereditary Melanoma Syndrome
  * Hereditary Pancreatic Syndrome
  * Li Fraumeni Syndrome
  * Cowden Syndrome
  * Hereditary Diffuse Gastric Cancer
  * Peutz Jeghers Syndrome
  * Juvenile Polyposis Syndrome
  * Ataxia Telangiectasia (Louis-Bar syndrome)

Individuals with a pretest mutation probability of > 2.5% based on validated published models 15

* Mismatch Repair (MMR)pro
* Prediction model for mutL homolog 1 (MLH1), muS homolg 2 (MSH2), and mutS homolog 6 (MSH6) gene mutations (Premm 1,2,6)
* Pancreas (Panc)Pro
* Melanoma (Mela)Pro
* Breast cancer (BRCA)Pro
* Breast and Ovarian Analysis of Disease Incidence and Carrier Estimation Algorithm (BOADICEA)
* International Breast Cancer Intervention Study (IBIS) (Tyler-Cuzick)
* Myriad II
* Phosphatase and tensin homolog (PTEN) Cleveland Clinic Score
* Clinical probability of > 2.5% where models are not available

Or one of the following:

Individuals with a phenotypic diagnosis of the following recognized cancer genetic syndromes which automatically confers a clinical chance of > 2.5%:

* Hereditary Breast and Ovarian Cancer
* Lynch Syndrome
* Familial or Attenuated Adenomatous Polyposis Syndrome
* Hereditary Melanoma Syndrome
* Hereditary Pancreatic Syndrome
* Li Fraumeni Syndrome
* Cowden Syndrome
* Hereditary Diffuse Gastric Cancer
* Peutz Jeghers Syndrome
* Juvenile Polyposis Syndrome
* Ataxia Telangiectasia (Louis-Bar syndrome) Participation will be open to patients of both sexes, all races and ethnic backgrounds, and of all ages. Subjects will include healthy individuals, cancer survivors, and patients actively being treated for cancer. Individuals at-risk for a hereditary cancer syndrome under age 18 will eligible for HCP testing if they meet the eligibility criteria with written parental consent and child assent where appropriate. Cognitively impaired adult subjects will be invited to participate through the written, informed consent of a legal representative designated on the consent form.

Exclusion Criteria:

Patients meeting one of the following criteria will be excluded the study

* Individuals with a pretest mutation probability of < 2.5% based on validated published models
* Prior genetic testing for germline cancer susceptibility
* Inability to provide written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: High-risk cancer genetics populations. Both male and female participants will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 1511 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Develop Hereditary Cancer panel repository | 3 years
  Develop a resource (repository and database) with banked specimens, HCP panel results, pre-clinical and follow up information and impact of the HCP results

SECONDARY OUTCOMES:
Analyze frequency of genes found on HCP panel in high-risk population | 3 years
  Summarize results of the HCP testing in terms of genes found with mutations and the frequency of mutation. The investigators will review expected versus actual off target or incidental findings from HCP testing. Off target findings will be classified into clinical actionable versus variants of uncertain significance (VUS). Incidence rates of off target mutations will be quantified and types of mutations will be qualitatively described.
Follow medical management of subjects after multi-gene panel testing | 5 years
  Summarize the medical management of these subjects - prior to testing after results disclosure of testing, and over the subsequent 5 years. The investigators will descriptively report changes to medical management from pre-cancer risk assessment and HCP testing and post-cancer risk assessment and HCP testing. For each patient, the investigators will determine whether the HCP result leads to a change in recommendation in regards to the risk reducing interventions and treatment.
Descriptive analysis of patient information gained through process | 5 years
  Perform descriptive analyses of information gained, in terms of reported patient experience and understanding of HCP testing. The investigators will measure the time it takes to reach a diagnosis with panel testing as compared to the sum of the average turnaround time (based on measurements supplied by Myriad Genetics) for sequential testing of single candidate genes. Bayesian models will be developed to measure the effect of an HCP actionable mutation result or an HCP VUS results on the final differential diagnosis of the patient. The Bayesian paradigm allows one to update the likelihood or probability of the event under consideration as more information becomes available.
  In addition to the questionnaire that subjects will complete about their intent to undergo risk-reducing interventions (Specific Aim 5), subjects will also complete a questionnaire to measure concerns and psychosocial issues associated with genetic testing.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Idos, MD, Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - University of Southern California/ Kenneth Norris, Jr. Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Stanford University, Stanford, California